CLINICAL TRIAL: NCT03961178
Title: Oncologic and Obstetric Outcomes After Conization for Uterine Cervical Lesion: A Cohort Study
Brief Title: A Cohort Study for the Following up of Conization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: CONE
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Precancerous Lesions; Conization; High Grade Intraepithelial Neoplasia; Uterine Cervical Cancer; Fertility; Pregnancy; Human Papillomavirus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: High-risk HPV — High-risk HPV testing for the cytology of lower genital tract
Diagnostic Test: TCT — Thin prep liquid-based cytology test for the cytology of lower genital tract

SUMMARY:
This study is to investigate the oncologic and obstetric outcomes in patients with conization for uterine cervical lesions from January 1, 2000 to January 1, 2019 in Peking Union Medical College Hospital.

The primary objectives consist of following:

1. The cumulative incidences of precancerous lesions and cancers of lower genital tract in patients who accepted conization for high grade intraepithelial neoplasia (HSIL), carcinoma in situ and stage IA1 cancer (FIGO 2009)
2. The cumulative pregnancy rates in patients sparing the fertility

The secondary objectives consist of following:

1. The effects of surgical protocols (modified Sturmdorf method and "8" figure suture) and energy equipment (cold knife and monopolar electrical cautery) on the oncologic and obstetric outcomes, and on the histological components.
2. A full description of histological components of the conization specimens
3. The cytological and virus outcomes after conization, based on the thin prep liquid-based cytology test (TCT) and high-risk human papillomavirus (HPV) testing

ELIGIBILITY:
Inclusion Criteria:

* Accepting conization in the study center
* Aged 18 years or older

Exclusion Criteria:

* Not meeting any of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients accepting conization in the study center who were aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-05-22 (Estimated); Study Completion 2021-05-22 (Estimated)

PRIMARY OUTCOMES:
The cumulative incidences of precancerous lesions or cancers | Five years
  The cumulative incidences of precancerous lesions and cancers of lower genital track in patients who accepted conization for high grade intraepithelial neoplasia (HSIL), carcinoma in situ and stage IA1 cancer (FIGO 2009)
The cumulative pregnancy rates | Five years
  The cumulative pregnancy rates in patients sparing the fertility

SECONDARY OUTCOMES:
The cytological results after conization | Five years
  The cytological after conization based on the thin prep liquid-based cytology test (TCT)
The virus outcomes after conization | Five years
  The virus outcomes after conization high-risk human papillomavirus (HPV) testing
The cumulative pregnancy loss rates | Five years
  The cumulative pregnancy loss rates in patients sparing the fertility
The cumulative live birth rates | Five years
  The cumulative live birth rates in patients sparing the fertility

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided